CLINICAL TRIAL: NCT02103907
Title: The Effect of Dynamic Balance Training on Balance and Physical Function in Those With Knee Osteoarthritis
Brief Title: Randomized Controlled Trial of Dynamic Balance Training in People With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Arthritis Health Professions Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H14-00587; AHPA-TAS- 14-001 (Other Grant/Funding Number: AHPA/The Arthritis Society)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Knee Osteoarthritis
Keywords: balance; knee; osteoarthritis; physical function
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait list (No Intervention): Wait list control group. Participants will be placed on the wait list and asked to maintain their current routine and level of activity during the 10 week period. Control group participants will receive the dynamic balance training program in a single training session after the followup (second testing session at 10 weeks).
- Treatment (balance training) (Experimental): Targeted dynamic balance training. Dynamic balance training will consist of progressive exercise training over three phases, with exercises emphasising dynamic balance control, muscle strength and proprioception. Exercises will be performed four times per week for ten weeks. Exercises will be taught and supervised by a trained kinesiologist. Difficulty of exercises will be increased progressively over time by increasing resistance, time of timed exercises, and distance of walking exercises. Exercises will be progressed to different exercises in each new phase (total 3 phases). Participants will complete six treatment sessions at the university (during weeks 1, 2, 3, 5, 7, and 9) that will be included in the total number of sessions per week. All other sessions will be performed at home.
  Interventions: Other: Targeted dynamic balance training

INTERVENTIONS:
Other: Targeted dynamic balance training — Participants in this study group will complete dynamic balance training exercises four times per week, for ten weeks. Exercise sessions at the university will last approximately one hour, and home exercise sessions will take approximately 30 minutes to complete. Exercises will emphasize dynamic balance control, muscle strength and proprioception and will be progressed over three phases during the ten weeks (with more difficult exercises phased in, and exercises that have been mastered phased out).
  Arms: Treatment (balance training)

SUMMARY:
There is a high prevalence of falls in those with knee osteoarthritis (OA) compared to healthy older adults. Balance is a key element of function that allows individuals to maintain posture and respond to perturbations, and poor balance control, a risk factor for falls, has been noted in those with knee OA. There is a lack of research guiding treatment for balance deficits in knee OA, with interventions aimed at improving balance deficits in those with knee OA having mixed results. Targeted dynamic balance interventions in other patient populations have been shown to significantly improve dynamic balance control and physical function. If results similar to such populations can be achieved, such a program may produce a significant reduction in functional disability in the knee OA population and improve quality of life. The purpose of this study is to examine the effect of a 10-week targeted dynamic balance intervention on dynamic balance and physical function in people with knee OA. This will be a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* age 50 - 80 years (to meet the American College of Rheumatology clinical definition of OA)
* radiographically confirmed knee OA in the medial compartment of the tibiofemoral joint
* predominance of pain/tenderness over the medial (inside) region of the knee

Exclusion Criteria:

* articular cartilage degradation in the lateral tibiofemoral compartment greater than the medial
* inflammatory arthritic condition
* history of knee or hip replacement surgery
* recent use of corticosteroids (oral or via injection, within last 6 months)
* pain originating predominantly from the patellofemoral joint
* inability to ambulate without a gait aid
* non-English speaking
* recent (within 6 months) arthroscopic knee surgery
* significant hip or back pain (limits the ability to perform the testing)
* Neurological, musculoskeletal or other condition that affects movement ability or balance (i.e. stroke, diabetes, Parkinson's, heart attack, multiple sclerosis, fibromyalgia)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in dynamic balance and mobility from baseline | 0, 10 weeks
  The Community Balance and Mobility Scale (CB&M) will be used to assess dynamic balance and mobility. The CB&M is a scale designed to assess dynamic balance and mobility and is administered by a trained assessor. The scale consists of 13 items including bending, walking, turning, and stair descent, with a maximum possible score of 96 and minimum score of 0. The scale has been validated and deemed reliable for use in the knee osteoarthritis population.
Change in self-reported physical function from baseline | 0, 10 weeks
  The Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) will be used to assess self-reported physical function. The WOMAC physical function subscale consists of 17 questions assessing physical function capabilities during activities of daily living.

SECONDARY OUTCOMES:
Change in knee pain from baseline | 0, 10 weeks
  Average pain over the previous week will be assessed using an 11-point numerical rating scale (0 = no pain; 10 = worst pain possible).
Change in fear of pain from baseline | 0, 10 weeks
  The Brief Fear of Movement Scale will be used to assess fear of pain. This scale is based on the widely used Tampa Scale of Kinesiophobia and contains 6 questions that evaluate fear of pain, movement and re-injury. The scale has been validated in individuals with OA.
Change in self-reported physical activity level from baseline | 0, 10 weeks
  The Physical Activity Scale for the Elderly score (PASE) will be used to measure self-reported physical activity level. This valid and reliable self-report instrument measures the type and level of recreational and occupational physical activity in the previous week.
Change in knee joint proprioception from baseline | 0, 10 weeks
  Knee joint proprioception will be measured using a knee joint repositioning task, previously used in those with OA to assess joint proprioception. Proprioception will be assessed in three randomly chosen target positions (15°, 30°, and 60° of knee flexion) while the participant is seated on an isokinetic dynamometer.
Change in muscle strength from baseline | 0, 10 weeks
  Maximal concentric and eccentric muscle strength of the plantarflexors, quadriceps, and hamstrings will be measured using the same isokinetic dynamometer as for the knee joint repositioning task.
Change in knee joint range of motion from baseline | 0, 10 weeks
  Range of motion will be measured using a goniometer, similar to other studies of knee OA. Participants will be asked to flex and extend their knee joint while supine.

OTHER OUTCOMES:
Ratio of number of exercise sessions attended to the maximum | 10 weeks
  Adherence to the exercise program will be assessed by calculating the number of exercise sessions attended divided by the maximum number of sessions.
Number of participants with adverse events | 10 weeks
  Adverse events experienced due to the intervention (i.e. increased knee pain) will be recorded weekly by participants.
Change in medication use | 10 weeks
  Any change in pharmacological use by participants will be recorded.
Change in co-interventions | 10 weeks
  Other therapies that participants may be pursuing will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Hunt, PT, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Motion Analysis and Biofeedback Laboratory, The University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Takacs J, Krowchuk NM, Garland SJ, Carpenter MG, Hunt MA. Dynamic Balance Training Improves Physical Function in Individuals With Knee Osteoarthritis: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1586-1593. doi: 10.1016/j.apmr.2017.01.029. Epub 2017 Mar 6. PMID 28279661